CLINICAL TRIAL: NCT00626691
Title: The Effects of Walnuts on Antioxidant Capacity and Nutritional Status in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: California Walnut Commission (Other); Tufts Medical Center (Other)
Responsible Party: Diane McKay, Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PV2707
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: antioxidant; walnut; nutritional status; Antioxidant capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Walnut consumption — Subjects will be randomized to receive either 0.75 oz (22.5 g) or 1.5 oz (45 g) of walnuts daily for the first 6 wk period, followed by a 6 wk washout period, and an additional 6 wk period during which they will receive the reverse dose of walnuts daily. Each serving of walnuts will be pre-weighed and pre-packaged.

SUMMARY:
The goal of this study is to find out if the daily consumption of English walnuts (Juglans regia L.) for 6 wk, at a dose readily incorporated into the diet (0.75 or 1.50 oz), will have a positive effect on antioxidant capacity and nutrient status in a population of healthy adults, aged 50-70 y.

DETAILED DESCRIPTION:
Epidemiological studies conducted in large populations have consistently shown that increased consumption of plant-based, antioxidant-rich foods, i.e., fruits, vegetables, grains, and nuts, reduces the risk for several chronic diseases. Among the various plants consumed worldwide, English walnuts (Juglans regia L.) have been reported to have the highest antioxidant activity, second only to rosehips (Rosa canina L.). There are a number of different compounds present in walnuts that are known to exhibit antioxidant activity, including vitamin E (as γ-tocopherol), melatonin, and several non-flavonoid polyphenols (e.g., ellagic acid monomers and polymeric ellagitannins). In vitro and ex vivo, studies have demonstrated the ability of walnuts and walnut extracts to increase the resistance of low density lipoprotein (LDL) to oxidation. Walnuts and/or their constituents have also been shown to decrease levels of oxidative stress in diabetic mice and increase serum antioxidant capacity in rats2. In humans, in vivo antioxidant capacity changes after consuming walnuts have only been measured in subjects with Type 2 diabetes. The antioxidant capacity of the lipophilic compartments, as well as the cooperative/synergistic interactions between the water- and fat-soluble antioxidants present in plasma after walnut consumption have not been measured. Indeed, there have been no studies conducted to date of the effect of walnut consumption on the total antioxidant capacity of healthy men and women. The goal of our proposed study is to determine if consuming walnuts in amounts readily incorporated into the diet can affect the antioxidant capacity of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and postmenopausal women age 50 or over
* BMI 18.5-35 kg/m2

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* History or known allergy to nuts of any kind
* Regular consumption of ≥ 5 oz nuts/week for 6 weeks prior to study admission
* Individuals taking estrogen
* Use of cholesterol-lowering medications
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 95 mmHg
* Regular use of oral steroids
* Regular daily intake of ≥ 2 alcoholic drinks
* Illicit drug use
* No fish oil supplements (including cod liver oil) for 6 weeks prior to study admission
* No high dose (≥ 3X RDA) supplements of vitamins C, E, selenium, or beta-carotene for one month prior to study admission
* No dietary supplements containing phenolic compounds, i.e., herbal preparations, or berry containing preparations (such as cranberry capsules) for one month prior to study admission
* No regular consumption of pomegranate juice (≥ 180 mL or 6 oz/d, ≥ 3 times/wk) for one month prior to study admission

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status and antioxidant capacity | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Diane L McKay, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] McKay DL, Chen CY, Yeum KJ, Matthan NR, Lichtenstein AH, Blumberg JB. Chronic and acute effects of walnuts on antioxidant capacity and nutritional status in humans: a randomized, cross-over pilot study. Nutr J. 2010 May 12;9:21. doi: 10.1186/1475-2891-9-21. PMID 20462428